CLINICAL TRIAL: NCT04685993
Title: An Open Label Extension Study of the Safety and Tolerability of LPCN 1144 for the Treatment of Subjects With Nonalcoholic Steatohepatitis (NASH) Who Have Completed the LPCN 1144-18-002 Trial
Brief Title: A Study of the Safety and Tolerability of LPCN 1144 in Subjects Who Completed the LPCN 1144-18-002 Trial
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Lipocine Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LPCN 1144-20-002
Record Dates: First submitted 2020-12-08; First posted 2020-12-28 (Actual); Results first posted 2024-07-17 (Actual); Last update posted 2024-07-17 (Actual); Status verified 2024-03

CONDITIONS: NASH - Nonalcoholic Steatohepatitis
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — testosterone undecanoate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment A (Experimental): LPCN 1144
  Interventions: Drug: LPCN 1144

INTERVENTIONS:
Drug: LPCN 1144 — Oral LPCN 1144, total daily dose of 450 mg testosterone undecanoate administered as BID (225 mg testosterone undecanoate per dose).
  Other Names: testosterone undecanoate

SUMMARY:
This is an open-label extension to Study LPCN 1144-18-002. The study is aimed at evaluating the safety and tolerability of LPCN 1144 in adult men with NASH.

DETAILED DESCRIPTION:
This is a multicenter, open-label extension protocol to provide LPCN 1144, an investigational drug, to subjects with NASH who have completed the LPCN 1144-18-002 protocol. Enrolled subjects will be given LPCN 1144 for up to 36 weeks. Subjects will be seen periodically to evaluate safety clinical laboratory tests, tolerability of LPCN 1144, adverse events, and overall subject health. Subjects will be given the option of having a liver biopsy performed at Week 36.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who have completed the 38 week study LPCN 1144-18-002 and wish to be treated with LPCN 1144
2. Subject must sign the Informed Consent Form to participate in the study

Exclusion Criteria:

1. Has participated or is participating in any other clinical (investigational) study after completion of LPCN 1144-18-002 study
2. Subjects who are currently receiving any androgens or estrogens
3. Subjects who are not willing to use adequate contraception for the duration of the study
4. Use of drugs historically associated with NAFLD (amiodarone, methotrexate, systemic glucocorticoids, tetracyclines, tamoxifen, estrogens, anabolic steroids, valproic acid, other known hepatotoxins) for more than 2 weeks in the 2 years prior to enrollment
5. Any other condition, which in the opinion of the investigator would impede compliance or hinder completion of the study

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2020-11-11 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2022-03-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anthony DelConte, Study Director — Lipocine Inc.
Locations (10):
- United States (10):
  - Clinical Trials Research, Roseville, California
  - Sensible Healthcare, LLC, Ocoee, Florida
  - Jubilee Clinical Research, Inc., Las Vegas, Nevada
  - R&H Clinical Research, Katy, Texas
  - Sun Research Institute, San Antonio, Texas
  - Endeavor Clinical Trials, San Antonio, Texas
  - Pioneer Research Soultions, Sugar Land, Texas
  - Advanced Clinical Research - Gut Whisperer, Riverton, Utah
  - Granger Medical Clinic, West Valley City, Utah
  - Manassas Clinical Research Center, Manassas, Virginia

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment A: LPCN 1144: Oral LPCN 1144, total daily dose of 450 mg testosterone undecanoate administered twice daily (225 mg testosterone undecanoate per dose).
Period: Overall Study
Arm/Group | Treatment A
Started | 25
Completed | 23
Not Completed | 2

BASELINE CHARACTERISTICS:
Population: Subjects who completed the 38 week study LPCN 1144-18-002 as planned and wanted to continue in this open label extension study
Arm/Group | Treatment A
Number analyzed (Participants) | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.8 (8.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9
  Not Hispanic or Latino | 16
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 24
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Safety and Tolerability of LPCN 1144
Description: Number of subjects presenting with a treatment-emergent adverse events
Time Frame: Baseline to Week 36
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment A
Number analyzed (Participants) | 25
Participants | 10

ADVERSE EVENTS:
Time Frame: 9 months
Arm/Group | Treatment A
All-Cause Mortality (participants affected / at risk) | 1/25
Serious Adverse Events (participants affected / at risk) | 1/25
Other Adverse Events (participants affected / at risk) | 2/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment A (N=25)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment A (N=25)
Upper respiratory infection (Infections and infestations) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After the multicenter publication or twelve months after the completion of the study, whichever occurs first, the PI may itself publish the results of its data from the study. The PI shall provide Sponsor with an advance copy of any proposed publication or oral presentation at least sixty days prior to the planned date of submission.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-02-01): https://cdn.clinicaltrials.gov/large-docs/93/NCT04685993/Prot_SAP_000.pdf